CLINICAL TRIAL: NCT04497467
Title: An Analysis of Changes in Out-patient Visits in Taiwan During the Time of Global COVID-19 Pandemic
Brief Title: Changes in Out-patient Visits in Taiwan During the Time of Global COVID-19 Pandemic
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202006225RINA
Record Dates: First submitted 2020-08-02; First posted 2020-08-04 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2023-10

CONDITIONS: Patient Preference
MeSH Terms: conditions — Patient Preference

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The COVID-19 pandemic becomes a global challenge. This study aims to analyze the possible changes in out-patient visits during the time of COVID-19 pandemic between January and June, 2020, compared with the same period in 2019, and the impact of the related healthy policies.

DETAILED DESCRIPTION:
Using the statistical data of the Health Insurance Bureau, this study aims to analyze the possible changes in out-patient visits during the time of COVID-19 pandemic between January and June, 2020, compared with the same period in 2019, and the impact of the related healthy policies.

ELIGIBILITY:
Inclusion Criteria:

* patients visited the out-patient clinic using the health insurance cards.

Exclusion Criteria:

* patients visited the out-patient clinic without using the health insurance cards.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: patients visited the out-patient clinic using the health insurance cards.
Sampling Method: Non-Probability Sample
Enrollment: 1200000 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
the number of the out-patient visits | 6 months
  Collect the number of the out-patient visits, comparing with that during the same period last year

CONTACTS AND LOCATIONS:
Overall Officials: Wan-Ching Lien, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan